CLINICAL TRIAL: NCT06759870
Title: 'Evaluation of the Effect of Increasing Surface Hydrophilicity by Photo-Functionalisation on Titanium Particle Release in Dental Implants by ICP-MS'
Brief Title: 'Evaluation of Photo-Functionalisation Effect on Dental Implants by ICP-MS'
Status: Not yet recruiting | Type: Observational
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Sukran Acipinar, Asst.Prof. Şükran ACIPINAR, Cumhuriyet University
Other Study IDs: Şükran Acıpınar ICP-MS; Cübap (Other Grant/Funding Number: Sivas Cumhuriyet University)
Record Dates: First submitted 2024-12-20; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Corrosion
Keywords: corrosion; dental implant; photo-functionalization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — saliva and gingival samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1- Standart dental implant
  Interventions: Other: Collection of saliva; Other: Collection of gingival samples; Other: ISQ registration
- 2-Photo-functionalization dental implant
  Interventions: Other: Collection of saliva; Other: Collection of gingival samples; Other: ISQ registration

INTERVENTIONS:
Other: Collection of saliva — An unstimulated saliva sample will be obtained for 1 minute before implant surgery and immediately after implant surgery.
Other: Collection of gingival samples — Gingival samples will be obtained by punch biopsy 3 months after implant surgery.
Other: ISQ registration — ISQ value will be record in placement dental implant.

SUMMARY:
Dental implants are used to rehabilitate and restore aesthetic and functional losses caused by tooth loss. They are made of titanium, which is considered to have the best biological safety as a material. However, it is known that implants can continuously corrode, releasing titanium particles and increasing the overall titanium content in the human body. This increased local concentration can lead to damage in intraepithelial hemostasis, exacerbation of inflammatory reactions in surrounding tissues, bone resorption, implant failure, allergic reactions, and accumulation in distal organs through blood and lymph pathways.

The surface properties of implants play a critical role in their corrosion behavior, with surface free energy and hydrophilicity providing advantages for implant osseointegration and wound healing. The titanium oxide layer covers the outer surface of the implant and helps maintain its integrity against external factors. It is known that UV light-mediated photo-functionalization reduces carbon concentration on the implant surface and increases oxygen levels, thereby improving the osseointegration of titanium. The hydroxylated oxide surface shows reactivity with ions, amino acids, and proteins in tissue fluid. Additionally, UV irradiation can create oxygen vacancies at bridging sites between titanium and oxygen atoms, forming a -OH hydrophilic layer in the outermost layer. Given that the oxide layer on the titanium surface provides corrosion resistance for implants, increasing surface hydrophilicity and thus strengthening osseointegration will also confer resistance to corrosion on titanium.

Although the mechanism of titanium particle release is not fully understood, it is influenced by the surface structure of the implant and wear from surgical operations, making it a concern that needs to be addressed.

In light of all this information, the aim of the study was to evaluate titanium particle release in implants with increased surface hydrophilicity by UV photofunctionalization during surgery and three months later during the healing process using ICP-MS.

DETAILED DESCRIPTION:
Nowadays, dental implants have become a common treatment for the removal of missing teeth. Studies on implant treatment have proven that titanium (Ti) implanted in bone continuously releases particles and significantly increases the total titanium content in the human body.

The two main reasons for the release of Ti particles from the implant are chemical corrosion and surface wear.

When the concentration of local titanium particles increases, oral intraepithelial haemostasis is damaged, inflammation in the surrounding tissues is exacerbated, and dynamic imbalance may occur in osteoblasts and osteoclasts . Ti ions and particles distributed in the human body are directly proportional to the distance from the implant. Concentration is higher in gingival and bone tissue adjacent to the implant.Recent publications in the dental implant literature have shown that treatment of dental implant titanium oxide (TiO) surfaces with 200-400 nm ultraviolet (UV) radiation can increase the bone-implant contact surface (BIC) after normal healing time. UV treatment induces energy to the surface electrons of TiO, and electron energy induces reactions to increase cell attachment and osteoblast contact. UV treatment acts mostly photochemically on titanium surfaces to increase hydrophilicity. UV treatment with this photo-functionalisation has been shown to increase biological reactivity and make the TiO surface attractive for cellular binding.

It has been shown that the hydrophilicity and electrical charge of the titanium surface play a key role in the initial attachment of cells to UV-treated titanium. The newly treated titanium surface is 'superhydrophilic'. This term is used when the contact angle of water to the surface is less than 5 degrees. Due to the ageing of titanium, the implant surface gradually becomes hydrophobic with a contact angle of more than 60 degrees after 4 weeks of treatment. However, it was observed that 5 minutes of UV exposure reduced the water contact angle to almost 0°. The main function of UV treatment is to change the surface from hydrophobic to superhydrophilic, with the removal of hydrocarbon contamination from the surface of titanium. This induced surface change increases the initial blood contact with the implant surface and facilitates cellular growth and osseointegration of bone to the implant. In fact, studies have shown that the bioactivity of UV-activated titanium surfaces is higher than the bioactivity of newly treated surfaces .

UV treatment of titanium surfaces increases the bone-implant contact area from 55% to close to 98.2% and also results in a 3-fold increase in the strength of bone-implant integration. This greatly improves primary stability even in implants placed without cortical bone support. Primary stability is very important to avoid micro-movements that may adversely affect the osseointegration process.

In the light of all this information, the aim of this study was to evaluate the effect of UV photo-functionalisation on titanium particle release in titanium implants.

ELIGIBILITY:
Inclusion Criteria:

* Standard size implant
* Non-smoker
* No other metal-containing restorations in the mouth

Exclusion Criteria:

* Soft or hard tissue augmentation
* Use of short implants or implants of 4.5 mm or more

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People between the ages of 35-65 who had dental implants and who did not have any systemic diseases constitute the population of our study.
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-02-03 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
ICP-MS (Inductively Coupled Plasma - Mass Spectrometer) results | 3 months
  The levels of titanium element will be measured on the ICP-MS device and the results will be expressed at ppb level.
ISQ (Implant stability quotient) result | 3 months
  ISQ values will be measured on the implant stability measurement device and expressed as numerical values.

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be uploaded to the system when the study is concluded.
Supporting Information: Study Protocol, SAP
Time Frame: Once the study is published, it is planned to remain in the system for 1 year.
Access Criteria: The study protocol may be made available publicly.